CLINICAL TRIAL: NCT06490575
Title: Using Nonpharmacological Approaches in Hypertension Prevention and Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Tandalayo Kidd, Professsor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10334
Record Dates: First submitted 2024-06-14; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: High Blood Pressure; Hypertension
Keywords: educational intervention; nonpharmacological approach; dietary behaviors; lifestyle behaviors
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The educational intervention was a randomized controlled trial in which participants were randomly divided into control and intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group received no educational or counseling sessions until the final post-survey questionnaires were administered.
- Nutrition Education (Experimental): Participants in the intervention group attended four face-to-face educational workshops (one session per week).
  Interventions: Other: Educational Intervention Based on Protection Motivation Theory to Improve Knowledge and Promote Nonpharmacological Approaches to Prevent and Manage Hypertension among Adults

INTERVENTIONS:
Other: Educational Intervention Based on Protection Motivation Theory to Improve Knowledge and Promote Nonpharmacological Approaches to Prevent and Manage Hypertension among Adults — Participants in the intervention group attended four face-to-face workshops (one session per week). Each session took about 30 minutes and consisted of lectures with PowerPoint presentations, discussion, questions and answers, and the distribution of educational pamphlets and booklets.
  Arms: Nutrition Education

SUMMARY:
The goal of this randomized controlled trial is to test the effectiveness of a four-module nutrition education resource promoting nonpharmacological approaches to prevent and manage hypertension. The main questions it aims to answer are:

* Does the educational intervention increase the knowledge of using nonpharmacological approaches in preventing and managing hypertension among participants?
* Does the educational intervention improve participants' lifestyle behaviors to prevent and manage hypertension? Researchers will compare a four-module educational intervention with a control group (no educational information received until after the study) to see if the educational intervention works to improve knowledge and healthy lifestyle behaviors in preventing and managing hypertension.

Participants will:

* Attend a 30-minute workshop every week for 4 weeks or no workshop at all
* Complete a survey on demographic information, knowledge, lifestyle behaviors, and quality of life at baseline and end of the study
* Complete a dietary 24-hour food recall at baseline, two weeks into the study, and at the end of the study
* Monitor blood pressure levels two times a day for four weeks

DETAILED DESCRIPTION:
Study Design:

This study is a randomized controlled trial with 30 participants randomly divided into control (n=15) and intervention (n=15) groups.

Pre- and post-survey Assessment:

All participants completed a comprehensive self-administered survey at baseline, which included:

* Knowledge related to hypertension and its management
* Lifestyle behaviors (diet, physical activity, alcohol intake, smoking status)
* Quality of life metrics
* Constructs from the Protection Motivation Theory (PMT), such as response efficacy, self-efficacy, perceived vulnerability, perceived severity, and intention

Dietary Assessment:

The Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) was used to assess participants' intake of fruits, vegetables, dietary sodium, and dietary potassium at three points:

* Baseline
* Mid-program (two weeks into the intervention)
* Post-intervention

Intervention:

The intervention group attended four weekly workshops, each lasting 30 minutes. The workshops were designed and led by a public health nutrition doctoral student and a nutrition expert. Each session included:

* Presentations with PowerPoint slides and interactive activities
* Group discussions
* Questions and answers
* Distribution of educational pamphlets and booklets

The educational sessions focused on:

* Increasing knowledge about hypertension prevention and management
* Promoting nonpharmacological approaches to prevent and manage hypertension, such as dietary changes and lifestyle modifications
* Addressing PMT components to influence participants' beliefs and intentions regarding their health behaviors

Control Group:

Participants in the control group did not receive any educational or counseling sessions during the intervention period. After the post-intervention survey, they were provided with all the educational materials and a brief overview of the contents.

Data Analysis:

Data collected from the surveys and ASA24 dietary assessments were analyzed using the Statistical Package for the Social Sciences (SPSS). Analyses focused on comparing changes in knowledge, lifestyle behaviors, quality of life, and dietary intake between the control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* currently residing in Riley County, Kansas
* a US citizen or a permanent resident
* proficient in English

Exclusion Criteria:

* younger than 18 years old
* neither a US citizen nor a permanent resident
* nonproficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Demographic and lifestyle pre- and post-survey instrument | 6 weeks
  The survey includes items on knowledge, risk perceptions, assessment of response efficacy and self-efficacy, intention for behavior change, and lifestyle behaviors.
ASA24 automated self-administered 24-hour food recall | 6 weeks
  This tool is based upon the validated Automated Multiple-Pass Method (AMPM) to collect dietary data using the 24-hour food recall.

SECONDARY OUTCOMES:
36-item quality of life | 6 weeks
  The SF-36 includes one multi-item scale that assesses four major components: general health, mental health, physical health, and social function.

CONTACTS AND LOCATIONS:
Overall Officials: Tandalayo Kidd, PhD, Principal Investigator — Kansas State University
Locations (1):
- Justin Hall, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Data are secured in a password-locked device. Only the researcher and the PI can access the research data due to confidentiality.

REFERENCES:
- [Result] Chatzinikolaou A, Tzikas S, Lavdaniti M. Assessment of Quality of Life in Patients With Cardiovascular Disease Using the SF-36, MacNew, and EQ-5D-5L Questionnaires. Cureus. 2021 Sep 14;13(9):e17982. doi: 10.7759/cureus.17982. eCollection 2021 Sep. PMID 34667665
- [Result] Carey RM, Whelton PK. The 2017 American College of Cardiology/American Heart Association Hypertension Guideline: A Resource for Practicing Clinicians. Ann Intern Med. 2018 Mar 6;168(5):359-360. doi: 10.7326/M18-0025. Epub 2018 Jan 23. No abstract available. PMID 29357396
- [Result] Schapira MM, Fletcher KE, Hayes A, Eastwood D, Patterson L, Ertl K, Whittle J. The development and validation of the hypertension evaluation of lifestyle and management knowledge scale. J Clin Hypertens (Greenwich). 2012 Jul;14(7):461-6. doi: 10.1111/j.1751-7176.2012.00619.x. Epub 2012 Apr 9. PMID 22747619
- [Result] Tsao CW, Aday AW, Almarzooq ZI, Anderson CAM, Arora P, Avery CL, Baker-Smith CM, Beaton AZ, Boehme AK, Buxton AE, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Fugar S, Generoso G, Heard DG, Hiremath S, Ho JE, Kalani R, Kazi DS, Ko D, Levine DA, Liu J, Ma J, Magnani JW, Michos ED, Mussolino ME, Navaneethan SD, Parikh NI, Poudel R, Rezk-Hanna M, Roth GA, Shah NS, St-Onge MP, Thacker EL, Virani SS, Voeks JH, Wang NY, Wong ND, Wong SS, Yaffe K, Martin SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2023 Update: A Report From the American Heart Association. Circulation. 2023 Feb 21;147(8):e93-e621. doi: 10.1161/CIR.0000000000001123. Epub 2023 Jan 25. PMID 36695182
- [Result] Carey RM, Whelton PK; 2017 ACC/AHA Hypertension Guideline Writing Committee. Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Synopsis of the 2017 American College of Cardiology/American Heart Association Hypertension Guideline. Ann Intern Med. 2018 Mar 6;168(5):351-358. doi: 10.7326/M17-3203. Epub 2018 Jan 23. PMID 29357392